CLINICAL TRIAL: NCT02640261
Title: Observational Prospective Study of the Success of Single Embryo Transfer Implantation Related to Level of Follicular Fluid Cytokines Expression in Low Responders Infertile Patients Treated With r-hLH add-on Therapy in a Second Controlled Ovarian Stimulation Cycle.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro di Procreazione Assistita Demetra (Other)
Responsible Party: Sponsor
Other Study IDs: Echelo
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2015-12

CONDITIONS: Female Infertility
Keywords: r-hLH; Cytokines; Follicular Fluid
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Follicular Fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Single embryo transfer on day 5, according to standard embryo morphological criteria
- Group 2: Single embryo transfer on day 5, chosen on the basis of both embryo morphological criteria and levels of cytokines measured in the individual FF.

SUMMARY:
The objective of our observational prospective study will be to compare, for women treated for infertility and included in a ICSI program, the implantation rate and delivery rate obtained after the transfer of a single blastocyst , chosen in a group of patients on the basis of the embryo morphology and in the other group on the basis of both embryo morphology and follicular fluid cytokines content.

100 IVF infertile patients , aged 32-39 years, with normal ovarian reserve, previously stimulated for their first cycle with standard short protocol (GnRH-Ant) and r-FSH alone, who have had a low ovarian response, Fort < 50% ( FORT Criteria, 2012; FORT= PFCX100/AFC), will be treated for the second cycle with standard short protocol (GnRH-Ant) and r-FSH plus r-LH , according to the standard established by our clinical practice.

Patients will be part of one of the following groups:

Group 1: single embryo transfer on day 5, according to standard embryo morphological criteria Group 2: single embryo transfer on day 5, chosen on the basis of both embryo morphological criteria and levels of cytokines measured in the individual FF.

ELIGIBILITY:
Inclusion Criteria:

* women age from < 38 years
* normal body mass index (BMI ) from 18 to 26
* parameters for ovarian reserve in the normal range (day 3 FSH levels < 10 mUI/ml ; day 3 E2 levels < 80 pg/ml; anti-mullerian hormone (AMH) levels > 1.5 ng/ml ; AFC (antral follicular count) > 6 )

Exclusion Criteria:

* polycystic ovary syndrome (PCOS)
* ovarian surgery
* pelvic endometriosis
* POR according to ESHRE criteria

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Normogonadotropic Infertile Women that failed the first IVFcycle and require r-hLh add on therapy as per Demetra clinical standard procedures
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 2 years

SECONDARY OUTCOMES:
Delivery Rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Chelo, MD, Principal Investigator — Clinica Center DEMETRA
Locations (1):
- DEMETRA, Florence, Italy, Italy